CLINICAL TRIAL: NCT05526508
Title: Use of Rebound Exercise in Community-dwelling Individuals With Neurological Disorders
Brief Title: Rebound Exercise in Neurological Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buckinghamshire New University (Other)
Responsible Party: Principal Investigator, Adaora Okemuo, Associate Lecturer, PhD research student, School of Health and Social Care Professions, Buckinghamshire New University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BNU2022Okemuo
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Neurological Diseases or Conditions
Keywords: neurological disorders; rebound; mini-trampoline; exercise /therapy; walking speed; fall risk; quality of life
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: There will be two frequency groups, once-weekly and twice-weekly, but the group's choice depends on the participants.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor will be blinded to the participant's frequency group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rebound once-weekly (Experimental): This group will undergo 12 weeks of rebound exercise training once weekly, for 30 minutes per session.
  Interventions: Device: Rebound exercise
- Rebound twice-weekly (Experimental): This group will undergo 12 weeks of rebound exercise training twice weekly, for 30 minutes per session.
  Interventions: Device: Rebound exercise

INTERVENTIONS:
Device: Rebound exercise — Exercise training on the rebounder/ mini-trampoline with stability handles attached

SUMMARY:
This study will be a pretest-posttest interventional trial investigating the use of rebound exercise in community-dwelling individuals with neurological disorders.

DETAILED DESCRIPTION:
Neurological disorders are linked to various problems, including but not limited to movement impairments, balance, fear of falls, reduced exercise tolerance, loss of muscle strength, reduced functional independence, sedentary behaviour and reduced quality of life. These impairments can lead to physical deconditioning, functional dependency and extreme disability if left unmanaged, creating the need for prompt treatment. Rebound exercise is an effective and safe form of aerobic exercise that has been successfully used in some populations. It can be included in rehabilitating people with neurological disorders for its beneficial effects on humans and minimal stress on the heart and joints. Its fun-giving experience makes it easier to engage regularly compared to traditional exercise tools that may feel like a task. It is also more affordable and less time-consuming than other standard modalities. The few available studies on rebound exercise in neurological disorders were mostly in inpatients, and evidence is scarce on the use of rebound exercise in community-dwelling individuals with neurological disorders. It is thus necessary to investigate its use in the community context as well as the minimal effective dosage of the intervention. This study will investigate the frequency of rebound exercise necessary to effect changes in physiological and functional outcomes such as heart rate, blood pressure, physical activity level, walking speed, risk of falls, cognitive function and quality of life. The enrolled participants will undergo 12 weeks of rebound exercise training once or twice weekly, depending on their frequency choice.

Ethical approval has been sought and obtained from the Research Ethics Committee of Buckinghamshire New University. Eligible volunteer participants will be asked to sign the informed consent after the study has been explained to them. They will be assured of data confidentiality by anonymising their information and will also be informed of their right to withdraw at any point.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a neurological disorder of upper motor neurone origin such as stroke, multiple sclerosis, Parkinson's disease, traumatic brain injury etc
* must score 3 or less on the Modified Rankin Scale for disability status
* must be able to walk with or without walking aids for at least 2 minutes
* have a body weight of <120 kg
* must be able to understand therapy instructions.

Exclusion Criteria:

* Pregnancy
* Other significant comorbidities
* cardiovascular or respiratory system disorders
* musculoskeletal disorders
* visual or auditory sensory disorders.
* cancer
* genu recurvatum

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in baseline risk of fall assessed by 3-Metre Backward Walk test at 12 weeks | Baseline and12 weeks
  3-metre backward walk test (3MBWT) is valid, reliable and clinically suitable to detect little changes in motor functions related to proprioception in patients with neurological diseases (Kocaman et al., 2021). Of all battery tests assessed for fall risks in patients with Parkinson's disease (Carter et al., 2020), 3MBWT had the highest overall accuracy for retrospective falls. Backward walking measures are more sensitive to identify age-related changes in mobility than forward walking. From a marked point, the patient is asked to walk backwards as fast and safely as possible to a 3-metre marked end. They are free to look back if they wish. A time of 3 seconds or less indicates good balance and low fall risk, while a time of 4.5 seconds or more indicates a high fall risk.
Change in baseline walking speed assessed by 10-Metre Walk test (10MWT) at 12 weeks | Baseline and 12 weeks
  10MWT has been shown to have excellent construct validity and reliability for patients with neurological diseases (Cheng et al., 2020). The individual is instructed to walk a set distance of 10 meters, and the time taken to walk the distance is noted. Assistive devices may be used but must be documented from test to test. Walking distance is measured in meters per second.
Change in baseline quality of life assessed by World Health Organisation Quality of Life Brief version (WHOQOLBREF) at 12 weeks | Baseline and12 weeks
  WHOQOLBREF is a 12-item questionnaire assessing physical and psychological domains of quality of life. The scale has been validated among stroke patients of different ethnic groups (Kerber et al., 2013; Post et al., 2011). It is rated on a 5-point Likert scale ranging from 1-5, with higher scores indicating better quality of life. A significant advantage it has over the more extended version is its reduced administration time (5 minutes), making it a more practical tool in research and clinical practice.
Change in baseline physical activity level assessed by International Physical Activity Questionnaire at 12 weeks | Baseline and 12 weeks
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients. The IPAQ can be used clinically and in population research that compares physical activity levels between populations internationally.
Change in baseline cognitive function assessed by mini-cog at 12 weeks | Baseline and 12 weeks
  The Mini-Cog is a simple screening test for cognitive impairment. It combines a brief memory test and a scored clock-drawing test. It allows rapid screening for short-term memory defects, learning and different cognitive abilities impaired in dementia patients.
Change in baseline blood pressure and heart rate assessed by digital blood pressure monitor at 12 weeks | Baseline and 12 weeks
  A digital Blood pressure monitor uses an inflatable air-bladder cuff, a battery-powered air pump and a pressure sensor for sensing arterial wall vibrations to measure blood pressure in an artery.

SECONDARY OUTCOMES:
Change in baseline grip strength assessed with a digital handheld dynamometer at 12 weeks | Baseline and 12 weeks
  A Hand-Held Dynamometer is a valid and reliable assessment tool used for objectively quantifying muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Yetunde M Dairo, PhD, Study Director — Buckinghamshire New University; Dearbhla Gallagher, PhD, Study Chair — Buckinghamshire New University
Locations (2):
- United Kingdom (2):
  - Buckinghamshire New University, Aylesbury, Buckinghamshire
  - Buckinghamshire New University, High Wycombe, Buckinghamshire

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data information necessary for publication of the study findings will be shared with the researchers
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Bhattacharya A, McCutcheon EP, Shvartz E, Greenleaf JE. Body acceleration distribution and O2 uptake in humans during running and jumping. J Appl Physiol Respir Environ Exerc Physiol. 1980 Nov;49(5):881-7. doi: 10.1152/jappl.1980.49.5.881. PMID 7429911
- [Background] Cugusi L, Manca A, Serpe R, Romita G, Bergamin M, Cadeddu C, Solla P, Mercuro G; Working Group of Gender Cardiovascular Disease of the Italian Society of Cardiology. Effects of a mini-trampoline rebounding exercise program on functional parameters, body composition and quality of life in overweight women. J Sports Med Phys Fitness. 2018 Mar;58(3):287-294. doi: 10.23736/S0022-4707.16.06588-9. Epub 2016 Jul 21. PMID 27441918
- [Background] Unver B, Sevik K, Yarar HA, Unver F, Karatosun V. Reliability of 3-m Backward Walk Test in Patients with Primary Total Knee Arthroplasty. J Knee Surg. 2020 Jun;33(6):589-592. doi: 10.1055/s-0039-1681099. Epub 2019 Mar 12. PMID 30861540
- [Background] Abit Kocaman A, Aydogan Arslan S, Ugurlu K, Katirci Kirmaci ZI, Keskin ED. Validity and Reliability of The 3-Meter Backward Walk Test in Individuals with Stroke. J Stroke Cerebrovasc Dis. 2021 Jan;30(1):105462. doi: 10.1016/j.jstrokecerebrovasdis.2020.105462. Epub 2020 Nov 13. PMID 33197801
- [Background] Cheng DK, Nelson M, Brooks D, Salbach NM. Validation of stroke-specific protocols for the 10-meter walk test and 6-minute walk test conducted using 15-meter and 30-meter walkways. Top Stroke Rehabil. 2020 May;27(4):251-261. doi: 10.1080/10749357.2019.1691815. Epub 2019 Nov 21. PMID 31752634
- [Background] Kerber KA, Brown DL, Skolarus LE, Morgenstern LB, Smith MA, Garcia NM, Lisabeth LD. Validation of the 12-item stroke-specific quality of life scale in a biethnic stroke population. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):1270-2. doi: 10.1016/j.jstrokecerebrovasdis.2012.08.011. Epub 2012 Sep 18. PMID 22995379
- [Background] Post MW, Boosman H, van Zandvoort MM, Passier PE, Rinkel GJ, Visser-Meily JM. Development and validation of a short version of the Stroke Specific Quality of Life Scale. J Neurol Neurosurg Psychiatry. 2011 Mar;82(3):283-6. doi: 10.1136/jnnp.2009.196394. Epub 2010 Aug 27. PMID 20802211
- [Background] Burandt P, Porcari JP, Cress ML, Doberstein S, Foster C, Green DJ (2016). ACE-Sponsored research: Putting mini-trampolines to the test. ACE Prosource. Available at www.acefitness.org Retrieved on 21/07/2022.
- [Background] Centers for Disease Control and Prevention (2022). Stroke statistics. CDC Wonder Online Database. Available at www.cdc.gov/stroke/facts Retrieved 21/07/2022
- [Background] Carter, V.A., Farley, B.G., Wing, K. and Jain, T.K., 2020. Diagnostic accuracy of the 3-meter backward walk test in persons with parkinson disease. Topics in Geriatric Rehabilitation, 36(3), pp.140-145